CLINICAL TRIAL: NCT04669938
Title: Role of the Microbiota in the Evolution of the SARS-CoV-2 Disease in Hospitalized Patients
Brief Title: Role of the Microbiota in the Evolution of the SARS-CoV-2 Disease,COVID-19, in Hospitalized Patients
Acronym: MicrobioCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201083
Record Dates: First submitted 2020-11-19; First posted 2020-12-17 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Gastrointestinal Microbiome; Viral Packaging Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized for COVID-19
  Interventions: Other: oropharyngeal and intestinal microbiota; Other: host genotype; Other: host immune factors; Other: viral sequence

INTERVENTIONS:
Other: oropharyngeal and intestinal microbiota — analysis of oropharyngeal and intestinal microbiota
Other: host genotype — analysis of a part of host genotype
Other: host immune factors — analysis of host immune factors
Other: viral sequence — analysis of viral sequence

SUMMARY:
Patients hospitalized for COVID-19 may need intensive care (e.g. mechanical ventilation) during hospitalization. Some risk factors are already known but better targeting of such patients is still needed, at least because existing risk factors are not strong enough to provide an accurate prediction. Care organization would benefit for such a predictive tool.

Oropharyngeal and gut microbiota could potentially fill a significant gap in predictive performances. The investigators therefore propose to sample 200 patients (oropharyngeal and rectal swab) admitted in infectious disease department at Bichat Hospital and at high risk of needing intensive care during hospitalization. The investigators plan to perform metagenomic sequencing and bioinformatic analysis of these samples to characterize the diversity of bacterial species present in the oropharynx and the gut and to identify new factors associated with the need for intensive care. Aside metagenomic analyses, The investigators will perform semi-quantitative cultures of the oropharyngeal and gut microbiota to identify and quantify pathogens in order to predict the risk of bacterial infections in COVD-19 patients.

For patients transferred in intensive care unit, The investigators will to perform another series of samples to better characterize the evolution of microbiota during mechanical ventilation and identify factors associated with the risk of developing a ventilator-associated pneumonia.

Microbiota data will be considered together with the host genotype, the viral sequence and a deep immunological profiling to identify the main determinants of the evolution toward severity of COVID-19.

DETAILED DESCRIPTION:
Patients hospitalized for COVID-19 may need intensive care (e.g. mechanical ventilation) during hospitalization. Some risk factors are already known (e.g. sex, comorbidities, initial clinical presentation inflammatory cytokines), but better targeting of such patients is still needed, at least because existing risk factors are not strong enough to provide an accurate prediction. Care organization would benefit for such a predictive tool.

Oropharyngeal and gut microbiota could fill a significant gap in predictive performances. The investigators therefore propose to take advantage of the French-COVID cohort and sample 200 patients (oropharyngeal and rectal swab) admitted in infectious disease department at Bichat Hospital and at high risk of needing intensive care during hospitalization. The investigators plan to perform metagenomic sequencing and bioinformatic analysis of these samples to characterize the diversity of bacterial species present in the oropharynx and the gut and to identify new factors associated with the need for intensive care. Aside metagenomic analyses, The investigators will perform semi-quantitative cultures of the oropharyngeal and gut microbiota to identify and quantify pathogens in order to predict the risk of bacterial infections in COVD-19 patients.

The genetic determinants of the host (the patient) could also be predictive of the severity of the disease and so does the immunological response to the COVID-19. Likewise, it has been suggested that certain mutations (notably the D614G mutation) of the viral sequence could be associated with the infectivity of the virus.

In addition to the direct role of the microbiota in the course of infection, the immune characteristics specific to the host, by themselves or in interaction with the microbiota, could play an important role in the progression of the disease.

This project focuses on the clinical characterization of COVID-19 and its evolution, as well as disease management.

The research focuses on 4 main areas:

* Characterization of the oropharyngeal and intestinal microbiota of patients with COVID-19
* Characteristics of the host (genotype)
* Immune characteristics of the host
* Characteristics of the SARS-CoV-2 viral genome

For patients transferred in intensive care unit, The investigators will to perform another series of samples to better characterize the evolution of microbiota during mechanical ventilation and identify factors associated with the risk of developing a ventilator-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with documented SARS-CoV-2 infection requiring hospitalization.

Exclusion Criteria:

* Lack of consent
* Patients hospitalized in an intensive care unit
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with documented SARS-CoV-2 infection requiring hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Identify risk factors associated with severe forms of COVID-19 requiring transfer to ICU | day 14
  The main endpoint is the indication of worsening of the general condition requiring transfer to ICU

SECONDARY OUTCOMES:
Link between the composition of the gut microbiota and admission to intensive care | 3 months
  Composition of the gut microbiota on admission to intensive care to predict the outcome of severe COVID-19 in patients transferred to the ICU (subgroup analysis)
Predictive performance of semi-quantitative culture and rapid metagenomic evaluation | 3 months
  Predictive performance of semi-quantitative culture and rapid metagenomic evaluation of the oropharyngeal microbiota to predict the occurrence of VAP in patients admitted to an ICU and mechanically ventilated (subgroup analysis).

CONTACTS AND LOCATIONS:
Locations (1):
- LESCURE, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided